CLINICAL TRIAL: NCT01335802
Title: Relation Between Thyroid Hormone Stimulated Mitochondrial Function and Spontaneous Abortion and Complications of Pregnancy in Subclinical Hypothyroidism
Brief Title: Relation Between Subclinical Hypothyroidism and Outcome of Pregnancy
Acronym: GravThyr
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne-Dorthe Feldthusen, MD, Naestved Hospital
Other Study IDs: SJ-177
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Abortion, Spontaneous; Pregnancy Complications; Subclinical Hypothyroidism
Keywords: Abortion, Spontaneous; Pre-eclampsia; Gestational hypertension; Pregnancy Complications; Subclinical hypothyroidism; Thyroperoxidase antibodies (TPOab); Mitochondrial dysfunction
MeSH Terms: conditions — Abortion, Spontaneous; Pregnancy Complications; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subclinical hypothyroidim: Women having subclinical hypothyroidism and/or TPOab-positive.
- Controls: Women having normal levels of TSH and TPOab-negative.

INTERVENTIONS:
Genetic:  — Genetic counseling

SUMMARY:
Studies have demonstrated a relationship between subclinical hypothyroidism and obstetrics complications like preterm delivery, pre-eclampsia, placental abruption and stillbirth. Subclinical hypothyroidism and positive thyroperoxidase antibodies (TPOab) may increase the risk of early spontaneous abortion before 12 weeks of gestation. But there is not a consensus if the prevalence of TPOab should be treated before and during pregnancy when the level of thyroid-stimulating hormone (TSH) is normal.

Thyroid hormones are regulators of the mitochondrial activity and our research group has previously shown that subclinical hypothyroidism affects mitochondrial activity.

The hypothesis:

Subclinical hypothyroidism causes early spontaneous abortion and or complications in pregnancy like pre-eclampsia because of mitochondrial dysfunction

DETAILED DESCRIPTION:
The aim is to estimate the relationship between SH and spontaneous abortion and/or obstetric complications because of mitochondrial dysfunction.

1. A prospective study where data from the General Suburban Population Study in Naestved will be analyzed to measure the frequency of subclinical hypothyroidism (SH) and TPOab. SH is defined as raised serum concentrations of TSH > 3,4 mU/l and normal levels of free T4 and T3. A cut-off of 60 mU/l is used for TPOab.
2. To estimate the relationship between SH or TPOab and early spontaneous abortion and pregnancy outcome. Inclusion of women who have experienced a minimum of one early spontaneous abortion and between 20 and 50 years old: 50 women who have SU and/or TPOab-positive and 50 women who have normal levels of TSH and TPOab-negative. The basal oxygen consumption will be measured and mitochondrial functions will be determined by flow cytometry.
3. To estimate the prevalence of gestational hypertension and pre-eclampsia among pregnant women with subclinical hypothyroidism and estimate the mitochondrial function. A minimum of 100 pregnant women without any thyroid disease or diabetes will be included.

Early spontaneous abortion is defined as abortion before 12 weeks of gestation. Obstetrics complications are defined as pre-eclampsia (proteinuria, oedema, hypertension), pregnancy-induced hypertension, placental insufficience (IUGR) and abruption, preterm delivery and stillbirth. Those complications will be analyzed from the data of the obstetric journals.

Measurement of oxygen consumption:

Respiratory gas analysis and volume measurements were performed with a canopy connected by a triple V (flow⁄gas sensor) to an Oxycon apparatus (Jaeger Oxycon Champion, Breda, the Netherlands). The equipment was calibrated before each test to compensate for ambient conditions such as air pressure, temperature and humidity. Basal VO2 was measured after at least 6 hours fasting. Before the test the individual resting pulse was established and the participants rested for about 30 min in a chair. The test room was quiet and the lighting was subdued. The subjects were given sufficient time to become familiarized with the equipment and the procedures and the test was initiated when the resting pulse was achieved. Oxygen consumption was measured when the uptake per minute remained constant. Measurements were performed for repeated periods of 30 seconds for 20 minutes. The method for recording oxygen uptake had a within-day variation of 0.8 % and a day-to-day variation of 5.8 %.

Measurement of mitochondrial mass (MM) and mitochondrial membrane potential (MMP) by flow cytometry:

Venous blood was drawn from the patient in EDTA Vacutainer tubes. From each patient 2 samples of 100 µl of blood were processed. One unstained control tube and one stained were analyzed.

The samples to be stained were added 1 µl Pacific Blue Mouse Anti-Human anti-CD14 (BD Biosciences, Denmark) and mixed. The tubes were incubated for 30 minutes at room temperature protected from direct light and subsequently washed.

The stained cells were resuspended in 890 µl PBS and added 10 µl 1 µM MTG (MitoTracker Green FM, Invitrogen A/S, Denmark) and 100 µl 1 µM TMRM (Tetramethylrhodamine methyl ester, Invitrogen A/S, Denmark). All stock solutions were dissolved in DMSO (dimethyl sulfoxide) and working solutions were diluted in PBS. After mixing samples were incubated for 30 minutes at room temperature in the dark.

ELIGIBILITY:
Part 2:

Inclusion Criteria:

Women who had experienced a minimum of one early spontaneous abortion and between 20 and 50 years old: 80 women who have subclinical hypothyroidism defined as raised serum concentrations of TSH > 3,4 mU/l and normal levels of free T4 and T3 or TPOab-positive and 80 women who have normal levels of TSH and TPOab-negative.

Exclusion Criteria:

* Women with metabolic disease, diabetes or psychiatric disease.
* Women using medicine against hypo- or hyperthyroidism.
* Women who never give birth or age more than 50 years.

Part 3:

Inclusion Criteria:

* Pregnant women (3rd trimester)

Exclusion Criteria:

* Women with metabolic disease, diabetes or psychiatric disease.
* Women using medicine against hypo- or hyperthyroidism.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Part 2: Fertile women from the General Suburban Population Study in Naestved (GeSuS), Region Zealand, Denmark.
  Part 3: Pregnant women (GA>27) who are consulting the department of obstetrics, Naestved Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-10; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Subclinical hypothyroidism | 1 year
  When the women participate the General Suburban Population Study (GeSuS) s-TSH are estimated. The women will be invited by letter if they match the inclusion criteria. There will only be one visit at the hospital for new bloodsample (flow cytometry) and measurement of oxygen consumption.
Pre-eclampsia | 1 year
  Does pregnant women with subclinical hypothyroidism have mitochondrial dysfunction which could explain the higher frequency of gestational hypertension and pre-eclampsia? Pregnant women who consult the department of obstetrics are invited to participate (interview and a blood sample).

SECONDARY OUTCOMES:
Mitochondrial dysfunction | 1 year
  Measure by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kvetny, MD, DMSc, Principal Investigator — Department of Internal Medicine & Faculty of Health Sciences, University of Copenhagen
Locations (1):
- Naestved Hospital, Næstved, Denmark